CLINICAL TRIAL: NCT06160297
Title: Investigation of the Effects of Modified Otago and Neuromuscular Exercise Programs on Falling, Gait, Physical Function and Quality of Life in Geriatric Knee Osteoarthritis
Brief Title: The Effects of Modified Otago and Neuromuscular Exercise on Falling and Physical Function in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Mehmet Ercan ODABAŞIOĞLU, PhD, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hkumeodabasioglu001
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; fall risk; modified Otago exercises; neuromuscular exercises; gait kinematics
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Modified Otago Exercise Group (Experimental): MOEG consists of strengthening and balance exercises. Participants were instructed to start the exercises with 5-minute flexibility exercises. The walking component of the original Otago exercises and the stair climbing exercise in the balance exercises were not included in the MOEG. The exercises included 5 strengthening exercises and 11 balance exercises.
  Interventions: Procedure: Modified Otago Exercise
- Neuromuscular Exercise Group (Experimental): Neuromuscular exercises basically consist of four exercise components. These; core stability / postural function, postural orientation, lower extremity muscle strength and functional exercises. Exercises also include 5-minute warm-up and cool-down periods.
  Interventions: Procedure: Neuromuscular Exercise
- Control Group (No Intervention): Traditional physiotherapy applications (Hotpack + US (Ultrasound) + TENS (Transcutaneous Electrical Stimulation) were applied to the control group initially, as in every group. After these applications, they were evaluated in terms of basic parameters. A re-evaluation was made after 12 weeks.

INTERVENTIONS:
Procedure: Modified Otago Exercise — The exercises are as follows;
  Warm-up exercises (5 min)
  Strengthening exercises (weight attached to ankle)
  * Knee extension while sitting on a chair
  * Knee flexion while standing with support from a chair
  * Hip abduction while standing with support from the chair
  Strengthening exercises (weight removed from ankle)
  * Standing on tiptoe with support from a chair
  * Rising on the heels with support from a standing chair
  Balance Exercises (progressively, with support - without support)
  * Mini squats
  * Toe walking
  * Walking on heels
  * Tandem stance
  * Tandem walking
  * Walking backwards (10 steps)
  * Standing on one leg
  * Assisted side walking
  * Side walking without support
  * Sit and stand on the chair
  * Figure eight walking
  Arms: Modified Otago Exercise Group
Procedure: Neuromuscular Exercise — * Proprioceptive stabilization of the knee with ball
  * Bridging with ball
  * Stepping forward, sideways and backwards by holding on to a fixed support while standing
  * Doing the same movements with the support leg on a different surface
  * Hip abduction-adduction with resistance band
  * Knee flexion-extension with resistance band
  * Climbing and descending steps by taking steps
  * Balancing on the step
  * Standing up from the chair
  Arms: Neuromuscular Exercise Group

SUMMARY:
. This study was carried out to examine the effects on walking, physical function and quality of life. There were 88 individuals in the study and they were divided into three groups as Modified Otago, Neuromuscular and Control groups. Traditional physiotherapy applications (Hotpack + Ultrasound (US) + Transcutaneous Electrical Nerve Stimulation (TENS) were applied to all groups. In addition to these applications, Modified Otago and Neuromuscular exercises were performed 2 days a week in a clinical setting, accompanied by a physiotherapist for 12 weeks. The control group was only followed up. Patients were evaluated for basic parameters before and after treatment: Berg Balance Scale (BBS) and Timed Up Go Test (TUG) for balance and fall risk, International Fall Efficiency Scale (FES-I) for fear of falling, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) for symptoms and function, Tampa Kinesiophobia Scale (TKS) for kinesiophobia, 6-minute walk test for functional capacity (6MWT), Nottingham Health Profile (NHP) for quality of life, McGill Short Form (MSF) questionnaire for pain, an android-based smartphone application called "Gait Analyzer" were used for spatio-temporal variables in gait. Joint position sense (JPS) was measured with a goniometer and knee flexion was determined as 30° and 60° target angles. The exercise experiences of the groups who exercised after the treatment were evaluated by asking three questions with answers ranging from 0 to 10. It was observed that modified Otago and Neuromuscular exercises reduced the risk of falling and fear of falling, increased balance, decreased clinical symptoms and pain, increased function and quality of life, provided positive changes in the spatio-temporal parameters of walking and partially improved the sense of joint position compared to the control group (p<0,05). When the exercise groups were compared, the Modified Otago group had more positive quality of life and pain than the Neuromuscular exercise group (p<0.05). In addition, individuals in this group evaluated the exercises as less boring and less tiring (p<0.001). Modified Otago and Neuromuscular exercises can be included in the treatment programs of individuals with geriatric knee osteoarthritis as exercises aimed at reducing possible falls. It was concluded that Modified Otago exercises are superior and therefore more preferable in terms of compliance and satisfaction of individuals.

DETAILED DESCRIPTION:
This study was conducted to geriatric individuals diagnosed with knee osteoarthritis who applied to T.R. Ministry of Health Kilis Prof. Dr. Alaeddin Yavaşca State Hospital Department of the Physical Therapy and Rehabilitation. 88 individuals who volunteered to participate in the study were included in the study. Individuals were evaluated in terms of basic parameters and 3 randomized groups were formed: Modified Otago exercise group (29), neuromuscular exercise group (29) and control group (30).

The study protocol was approved by Hasan Kalyoncu University Ethics Committee (No: 2021/073, 31.05.2021). Individuals were informed about the scope, duration, treatment and evaluations of the study.

The study was planned as prospective, single-blind and randomized controlled. Patients underwent a preliminary evaluation by a physiotherapist to determine compliance with the inclusion criteria. The numbers were randomly distributed on the website www.random.org, which offers random numbers for many purposes. Patients whose eligibility was determined were then assigned to one of these groups in the order of arrival. The groups were determined as Group-1 Modified Otago Exercise Group (MOEG), Group-2 Neuromuscular Exercise Group (NEG) and Group-3 Control Group (CG).

Initially, traditional physiotherapy applications (Hotpack + US (Ultrasound) + TENS (Transcutaneous Electrical Stimulation) were applied to each group, and after these applications, each group was evaluated in terms of basic parameters.

In addition to these practices, the exercise groups were given modified otago and neuromuscular exercises in the clinic, 2 days a week, under the supervision of a physiotherapist, for 12 weeks. KG was not intervened.

Patients were evaluated for basic parameters before and after treatment. Berg Balance Scale (BBS) and Timed Up and Go Test (TUG) for balance and fall risk in individuals, International Fall Activity Scale (FES-I) for fear of falling, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) for disease-specific symptoms and functional status, Tampa Kinesiophobia Scale (TKS) for kinesiophobia, 6-minute walk test (6MWT) for functional capacity, Nottingham Health Profile (NHP) for quality of life, McGill Short Form (MSF) questionnaire for pain, "Gait Analyzer" for spatio-temporal variables of gait that an android-based smartphone application called was used. For joint position sense (EPH), 30° and 60° knee flexion were determined as target angles and measurements were made with a goniometer.

At the end of 12 weeks, all groups were re-evaluated in terms of basic parameters.

Functional Status Assessment: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a self-reported health status measure developed to assess pain, joint stiffness, and function that is widely used in patients with hip and knee osteoarthritis. It questions patients clinically about three different dimensions: pain, joint stiffness and function in the last 24 hours. Questions are in a 5-point Likert format and are scored between 0-4 (0: none, 1: mild, 2: moderate, 3: severe, 4: very severe). It contains a total of 24 questions: 5 assessing pain, 2 assessing stiffness, and 17 assessing function. The three subscales that make up the scale can be scored separately or as a total. Higher scores represent worse pain, physical function, and stiffness.

Balance and Fall Risk Assessment:

Berg Balance Scale (BBS): BBS is used to evaluate an adult's balance abilities while performing functional tasks. Some functional activities such as standing up from a sitting position, standing without support, standing on one leg, various turning activities, standing with eyes closed, and chair transfers are evaluated. The scale consists of 14 items in Likert format and performances are scored as five different points (0-4), ranging from 0 "cannot do" to 4 "does independently and safely". The total score is between 0 and 56 points. The closer this value is to 0, the higher the risk of falling. According to the total score obtained from this test, if the risk of falling is between 0-20 points, it is considered as "high risk", if it is between 21-40 points, it is considered as "medium risk", and if it is between 41-56 points, it is considered as "low risk". Patients with moderate fall risk were included in our study.

Timed Up and Go Test (TUG): Recommended by the American Geriatrics Society and the British Geriatrics Society to screen for fall risk. This test was used to determine functional mobility and fall risk. For the test, patients were asked to sit on a chair. A target point was determined 3 meters away from the chair. Patients were instructed to stand up, walk to this target at a steady and normal walking speed, then return and sit on the chair. The time between the patients getting up from the chair and sitting back down was measured with a stopwatch. The patients made the first trial for learning and the second trial was recorded in seconds as the real test.

Assessment of Fear of Falling: (Falls Efficacy Scale - International FES-I): International Falls Efficacy Scale is a 16-question self-reported scale that aims to obtain information about individuals' anxiety levels regarding falls while performing daily life activities. The questions are in Likert format and are scored as 4 points (1-4), from 1 "I am not worried at all" to 4 "I am very worried". The total score varies between 16-64 points, and the closer this score is to 64, the higher the fear of falling.

Assessment of Kinesiophobia: Kinesiophobia is a condition in which a patient has an excessive, irrational, and debilitating fear of physical activity and movement resulting from a painful injury or a feeling of vulnerability to re-injury. To evaluate individuals' kinesiophobia, the Tampa Kinesiophobia Scale, whose Turkish reliability and validity has been established, was used. The scale is in a four-point Likert format (1-totally disagree, 4-totally agree) and consists of 17 questions. While calculating the scale score, the scores of some questions (4, 8, 12 and 16) are reversed and calculated. A high total score indicates that the individual has high kinesiophobia.

Functional Capacity Evaluation: Functional capacity evaluation of individuals was carried out with the 6-minute walk test (6MWT). 6MWT not only evaluates the patient's walking ability but also gives an indication of the individual's endurance level. Therefore, it is an excellent functional outcome measure for knee OA recommended by the ACR. The test is performed in a closed and uncrowded place. In a closed area, there should be a flat surface with a distance of 30 meters between the starting and ending points. The distance an individual can walk in this area in 6 minutes is evaluated in meters. Before the test begins, the patient is rested and given information about the test. The patient is asked to walk at his own walking pace between the starting and ending points. The test is monitored with a stopwatch. The purpose of the test is to measure the maximum distance he can walk during this time.

Assessment of Pain: Pain status of individuals was evaluated with the Turkish version of the short form McGill pain questionnaire. The questionnaire consists of three parts and provides information about the sensory, emotional and intensity component of pain sensation. In the first section, there are 15 different words describing pain, and there are options in a four-point Likert format (0-none, 1-mild, 2-moderate, 3-severe) corresponding to the intensity of the defined pain level. The individual is asked to indicate the type and intensity of pain he is experiencing. The first 11 questions evaluate the sensory dimension of pain and the last 4 questions evaluate the perceptual dimension of pain. In the first part, three different scores are obtained: sensory pain score, perceptual pain score and total pain score. In the second part of the questionnaire, there are six different expressions ranging from "none" to "unbearable pain" to determine the severity of the current pain experienced by the individual. In the third part, there is a visual pain scale in the form of a line divided into 1 cm slices to determine the severity of the individual's current pain (no pain - 0, severe pain - 10). The individual is asked to indicate the intensity of pain he/she experiences as requested in the second and third sections. With the third part, a visual pain score is obtained.

Evaluation of Quality of Life: The Turkish version of the Nottingham Health Profile (NHP) was used to evaluate individuals' perceptions of quality of life. NHP is a quality of life scale used to measure individuals' perceived health status. It has been found to be extremely safe for use in OA populations. The survey essentially consists of two parts. The first part deals with 6 health-related dimensions (pain-8, physical activity-8, energy level-3, sleep-5, social isolation-5 and emotional reactions-9) and consists of a total of 38 items. The second part consists of 7 items. Individuals are asked to evaluate the situations as "yes" or "no". Each section is scored between 0-100 points and the total score is scored between 0-600 points, thus obtaining a health profile score. Low scores indicate a good health profile, high scores indicate a poor health profile.

Joint Position Sense: Joint position sense (JPS) is evaluated by the angular difference between a repeatedly determined target position and the predicted position, and this is called absolute angular error. This method is a reliable technique for the knee joint. JPS is tested by actively finding the joint position that was previously taught passively. In the study, only the knee joint was evaluated for JPS and 30° and 60° knee flexion were determined as target angles. A universal goniometer was used for testing. Before the measurement, individuals were given information about the test. For the test position, individuals were placed in a sitting position with their hips and knees flexed at 90° and their feet elevated from the ground. Then, while the knee was slowly brought from 90° flexion to passive extension, it was first stopped at 60° flexion angle for 5 seconds and the individuals were asked to perceive and learn this position. Then, the measurement was made by asking the individual to bring his knee to this target angle. The difference was recorded as absolute angular error. The same process was performed for the 30° flexion angle. Three repetitions were requested for both positions and the averages were calculated and recorded. Individuals used an eye patch to eliminate visual feedback while testing.

Evaluation of Spatio-Temporal Variables of Gait: For gait, a smartphone-based application called "Gait Analyzer" for gait (version 0.9.95.0 (Control One LLC, NM, USA)), offered as a paid application by the Android platform, whose reliability and validity have been tested-retested, was used. As a result of the measurement made with this application, kinematic data of walking such as walking speed, cadence, step time, step length, step length symmetry and step time symmetry can be obtained. After the program was installed on the smartphone (Huawei Mate 10 Lite, RNE-L01), some demographic data of the patient was entered. Afterwards, the smartphone was fixed to the area corresponding to the patient's L3 proccesus spinosus with a suitable waist belt with a velcro bandage. The measurement was then performed by asking the patients to walk a distance of 20 meters in their natural walking style and speed, without walking aid. The results were recorded on the form.

Assessing Exercise Satisfaction: A form with numerical scores between 0-10 was applied to the Modified Otago and Neuromuscular exercise group at the end of 12 weeks for their exercise experiences. The form included the following 3 questions: "Were you satisfied with the treatment?", "Did you have difficulty doing the exercises?" and "Did you get bored doing the exercises?".

Exercise Protocols: For both exercise models, before starting the intervention, individuals were informed about the exercise procedures and shown in detail how to do the exercises. They were informed that the movements should be performed correctly while the exercises were performed, that the exercises should be accompanied by the correct breathing pattern, and that they could rest if they felt tired. She was told to report any shortness of breath, dizziness, or chest pain during exercise to the physiotherapist. The exercises took approximately 20 minutes to complete and were performed 2 non-consecutive days a week in a clinical environment, accompanied by a physiotherapist. Individuals were assigned two days a week for exercise sessions. A make-up option was offered the same week for the days he could not attend the session. Individuals whose participation in the program was below 75% were excluded from the study.

Modified Otago Exercise Group (MOEG) MOEG consists of strengthening and balance exercises. Participants were instructed to start the exercises with 5-minute flexibility exercises. The walking component of the original Otago exercises and the stair climbing exercise in the balance exercises were not included in the MOEG. The exercises included 5 strengthening exercises and 11 balance exercises.

There are basically four difficulty levels in Otago exercises: A, B, C and D, from easy to difficult. But not every exercise involves these four levels. While some exercises are performed at a single difficulty level, some may include all four levels in the process. While the exercises were performed, progression was made according to the individuals' ability to achieve these difficulty levels. In general, if individuals could perform 2 sets of 10 repetitions at a difficulty level with quality, they were moved to a higher difficulty level. In the first two weeks of the intervention, the exercises were started from the simplest level for all individuals so that the individuals could learn the exercises more easily and adapt to the program.

A 1 kg free weight attached to the ankle was used as resistance in the strengthening exercises of knee extension, knee flexion and hip abduction. In the first two weeks of the intervention, all individuals started with 1 kg. When the movements were performed with quality in 2 sets of 10 repetitions, the free weight was increased to 2 kg and continued in this way for the remaining weeks. Body weight was used as resistance in dorsiflexor and plantar flexor strengthening exercises. There were two difficulty levels in these exercises: supported and unsupported. The progression continued in the same way, when the movements were performed in 2 sets of 10 repetitions with high quality, they moved to a higher difficulty level and continued at this level for the remaining weeks. In balance exercises, progression was made by first moving from the supported position to the unsupported position, and then by increasing the number of repetitions. When the movements were performed in a quality manner for 2 sets of 10 repetitions, the movements were continued to a higher difficulty level, as in the strengthening exercises.

The exercises are as follows; Warm-up exercises (5 min) Strengthening exercises (weight attached to ankle)

* Knee extension while sitting on a chair
* Knee flexion while standing with support from a chair
* Hip abduction while standing with support from the chair Strengthening exercises (weight removed from ankle)
* Standing on tiptoe with support from a chair
* Rising on the heels with support from a standing chair Balance Exercises (progressively, with support - without support)
* Mini squats
* Toe walking
* Walking on heels
* Tandem stance
* Tandem walking
* Walking backwards (10 steps)
* Standing on one leg
* Assisted side walking
* Side walking without support
* Sit and stand on the chair
* Figure eight walking Neuromuscular Exercise Program Neuromuscular exercises basically consist of four exercise components. These; core stability / postural function, postural orientation, lower extremity muscle strength and functional exercises. Exercises also include 5-minute warm-up and cool-down periods. Progression in neuromuscular exercises was achieved by changing the direction and speed of the movement from simple to difficult according to the capacities of the individuals, increasing the amount of loading, changing the support surface and perturbation interventions. Apart from this, the resistance bands used in strengthening exercises started with yellow color and were switched to red, green and purple colors in the following weeks, depending on the capacity of the individual. In general, if individuals could perform 2 sets of 10 repetitions at a difficulty level with quality, they were moved to a higher difficulty level. In the first two weeks of the intervention, the exercises were started from the simplest level for all individuals so that the individuals could learn the exercises more easily and adapt to the program.
* Proprioceptive stabilization of the knee with ball
* Bridging with ball
* Stepping forward, sideways and backwards by holding on to a fixed support while standing
* Doing the same movements with the support leg on a different surface
* Hip abduction-adduction with resistance band
* Knee flexion-extension with resistance band
* Climbing and descending steps by taking steps
* Balancing on the step
* Standing up from the chair

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee OA
* 65 years and above - 80 years and below
* BMI <30 kg/m2
* 3 < VAS score < 8
* Berg Balance Scale scores between 21-40
* Have a score of 24 or above on the Standardized Mini Mental State Test
* Not having received physiotherapy treatment in the last year.
* Able to adapt to the training program,
* Those who want to participate in volunteer work,
* Individuals with informed consent

Exclusion Criteria:

* Patients with positive Romberg Test
* Patients with absolute angular error value more than 20˚ in the evaluation of joint position sense
* Patients with B12 deficiency
* Patients using antidepressant, anxiolytic and myorelaxant derivative drugs
* Patients diagnosed with diabetes
* Patients with discopathy
* Those who have had lower extremity surgery, traumatic injury within the last six months, or are currently involved in a rehabilitation program
* Refusing to participate in the study
* Patients who cannot adapt to the training program.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Functional Status Assessment | 3 months
  WOMAC is a self-reported health status measure developed to assess pain, joint stiffness, and function that is widely used in patients with hip and knee osteoarthritis.
Fall Risk Assessment | 3 months
  Berg Balance Scale (BBS): BBS is used to evaluate an adult's balance abilities while performing functional tasks. Some functional activities such as standing up from a sitting position, standing without support, standing on one leg, various turning activities, standing with eyes closed, and chair transfers are evaluated. The scale consists of 14 items in Likert format and performances are scored as five different points (0-4), ranging from 0 "cannot do" to 4 "does independently and safely". The total score is between 0 and 56 points. The closer this value is to 0, the higher the risk of falling.
Balance Assessment | 3 months
  Timed Up and Go Test (TUG) :Recommended by the American Geriatrics Society and the British Geriatrics Society to screen for fall risk. This test was used to determine functional mobility and fall risk. For the test, patients were asked to sit on a chair. A target point was determined 3 meters away from the chair.
Assessment of Fear of Falling | 3 months
  Falls Efficacy Scale - International FES-I :International Falls Efficacy Scale is a 16-question self-reported scale that aims to obtain information about individuals' anxiety levels regarding falls while performing daily life activities. The questions are in Likert format and are scored as 4 points (1-4), from 1 "I am not worried at all" to 4 "I am very worried". The total score varies between 16-64 points, and the closer this score is to 64, the higher the fear of falling.
Spatio-Temporal Variables of Gait | 3 months
  For gait, a smartphone-based application called "Gait Analyzer" for gait (version 0.9.95.0 (Control One LLC, NM, USA)), offered as a paid application by the Android platform, whose reliability and validity have been tested-retested, was used. As a result of the measurement made with this application, kinematic data of walking such as walking speed, cadence, step time, step length, step length symmetry and step time symmetry can be obtained. After the program was installed on the smartphone (Huawei Mate 10 Lite, RNE-L01), some demographic data of the patient was entered. Afterwards, the smartphone was fixed to the area corresponding to the patient's L3 proccesus spinosus with a suitable waist belt with a velcro bandage. The measurement was then performed by asking the patients to walk a distance of 20 meters in their natural walking style and speed, without walking aid. The results were recorded on the form.
Evaluation Quality of Life | 3 months
  The Turkish version of the Nottingham Health Profile (NHP) was used to evaluate individuals' perceptions of quality of life. NHP is a quality of life scale used to measure individuals' perceived health status. It has been found to be extremely safe for use in OA populations. Turkish adaptation and psychometric properties study of the questionnaire was conducted by Küçükdeveci et al. It was conducted by in individuals with OA. The survey essentially consists of two parts. The first part deals with 6 health-related dimensions (pain-8, physical activity-8, energy level-3, sleep-5, social isolation-5 and emotional reactions-9) and consists of a total of 38 items. The second part consists of 7 items. Individuals are asked to evaluate the situations as "yes" or "no". Each section is scored between 0-100 points and the total score is scored between 0-600 points, thus obtaining a health profile score. Low scores indicate a good health profile, high scores indicate a poor health profile.

SECONDARY OUTCOMES:
Pain Assessment | 3 months
  Pain status of individuals was evaluated with the Turkish version of the short form McGill pain questionnaire. The questionnaire consists of three parts and provides information about the sensory, emotional and intensity component of pain sensation. In the first section, there are 15 different words describing pain, and there are options in a four-point Likert format (0-none, 1-mild, 2-moderate, 3-severe) corresponding to the intensity of the defined pain level.
Functional Capacity Evaluation | 3 months
  Functional capacity evaluation of individuals was carried out with the 6-minute walk test (6MWT). 6MWT not only evaluates the patient's walking ability but also gives an indication of the individual's endurance level. Therefore, it is an excellent functional outcome measure for knee OA recommended by the ACR.
Assessing Exercise Satisfaction | 3 months
  A form with numerical scores between 0-10 was applied to the Modified Otago and Neuromuscular exercise group at the end of 12 weeks for their exercise experiences. The form included the following 3 questions: "Were you satisfied with the treatment?", "Did you have difficulty doing the exercises?" and "Did you get bored doing the exercises?".
Assessment of Kinesiophobia | 3 months
  Kinesiophobia is a condition in which a patient has an excessive, irrational, and debilitating fear of physical activity and movement resulting from a painful injury or a feeling of vulnerability to re-injury. To evaluate individuals' kinesiophobia, the Tampa Kinesiophobia Scale, whose Turkish reliability and validity has been established, was used. The scale is in a four-point Likert format (1-totally disagree, 4-totally agree) and consists of 17 questions. While calculating the scale score, the scores of some questions (4, 8, 12 and 16) are reversed and calculated. A high total score indicates that the individual has high kinesiophobia.
Joint Position Sense | 3 months
  Joint position sense (JPS) is evaluated by the angular difference between a repeatedly determined target position and the predicted position, and this is called absolute angular error. This method is a reliable technique for the knee joint. JPS is tested by actively finding the joint position that was previously taught passively. In the study, only the knee joint was evaluated for JPS and 30° and 60° knee flexion were determined as target angles. A universal goniometer was used for testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided